CLINICAL TRIAL: NCT07244965
Title: Neoadjuvant Ivonescimab Combined With Paclitaxel and Cisplatin, Followed by Concurrent Chemoradiotherapy in Patients With High-Risk Locally Advanced Cervical Cancer：A Phase II, Single-Arm Study
Brief Title: Neoadjuvant Ivonescimab Plus Chemotherapy Followed by Concurrent Chemoradiotherapy in High-Risk Locally Advanced Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO2024-752
Record Dates: First submitted 2025-08-25; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-06

CONDITIONS: LOCALLY ADVANCED CERVICAL CANCERS
Keywords: Ivonescimab; Cervical Cancer; Neoadjuvant; Immune Checkpoint Inhibitor; Concurrent Chemoradiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Drug Therapy; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Ivonescimab Plus Paclitaxel and Cisplatin, Followed by Chemoradiotherapy (Experimental): Participants in this arm will receive two cycles of neoadjuvant therapy consisting of Ivonescimab (20 mg/kg, intravenous infusion on Day 1 of each 21-day cycle) combined with paclitaxel (175 mg/m² or albumin-bound paclitaxel 260 mg/m²) and either cisplatin (75 mg/m²) or carboplatin (AUC = 5), at the discretion of the investigator. After completion of neoadjuvant treatment, participants will undergo concurrent chemoradiotherapy with weekly cisplatin (40 mg/m² × 5 weeks) or carboplatin (AUC = 2), in combination with pelvic external beam radiation therapy (EBRT) and brachytherapy per institutional protocol.
  Interventions: Drug: Ivonescimab Combined With Chemotherapy; Combination Product: CONCURRENT CHEMORADIATION (CISPLATIN)

INTERVENTIONS:
Drug: Ivonescimab Combined With Chemotherapy — Participants will receive neoadjuvant therapy consisting of Ivonescimab at 20 mg/kg administered via intravenous infusion on Day 1 of each 21-day cycle, for a total of 2 cycles. Ivonescimab will be administered in combination with paclitaxel (175 mg/m², intravenous infusion) or albumin-bound paclitaxel (260 mg/m², intravenous infusion), and cisplatin (75 mg/m², intravenous infusion) or carboplatin (AUC = 5). All chemotherapy drugs are administered on Day 1 of each cycle. The choice between cisplatin or carboplatin, and between solvent-based or albumin-bound paclitaxel, will be made at the investigator's discretion based on patient tolerance and clinical condition.
Combination Product: CONCURRENT CHEMORADIATION (CISPLATIN) — Following completion of neoadjuvant therapy, participants will undergo concurrent chemoradiotherapy consisting of weekly cisplatin (40 mg/m², intravenous infusion, once per week for 5 weeks) or carboplatin (AUC = 2, once weekly for 5 weeks), administered concurrently with pelvic external beam radiation therapy (EBRT) and intracavitary brachytherapy. Radiotherapy will be delivered per institutional standards, including a total pelvic EBRT dose of approximately 45-50.4 Gy in 25-28 fractions and image-guided brachytherapy with a total equivalent dose of at least 80-85 Gy EQD2 to point A or tumor residual volume. The choice of chemotherapy agent and radiation technique will be determined by the investigator based on clinical condition and institutional protocol.

SUMMARY:
This is a single-arm, phase II clinical trial evaluating the efficacy and safety of neoadjuvant Ivonescimab combined with paclitaxel and cisplatin (TP regimen), followed by concurrent chemoradiotherapy, in patients with high-risk, locally advanced cervical cancer (FIGO stage III-IVA). Eligible participants will receive two cycles of neoadjuvant Ivonescimab plus TP chemotherapy, followed by standard concurrent chemoradiotherapy. The primary endpoints include progression-free survival (PFS) and objective response rate (ORR) following neoadjuvant treatment. Secondary endpoints include overall survival (OS), disease control rate (DCR), safety, and quality of life (EORTC QLQ-C30). Exploratory analysis will focus on identifying predictive biomarkers for Ivonescimab efficacy.

DETAILED DESCRIPTION:
This is an open-label, single-arm, phase II clinical trial designed to evaluate the efficacy and safety of neoadjuvant Ivonescimab combined with paclitaxel and cisplatin (TP regimen), followed by concurrent chemoradiotherapy, in patients with high-risk, locally advanced cervical cancer (FIGO 2018 stage III-IVA) who are not candidates for radical surgery.

Eligible patients will receive two cycles of neoadjuvant therapy consisting of Ivonescimab (20 mg/kg, intravenous infusion on day 1) plus paclitaxel (175 mg/m² or albumin-bound paclitaxel 260 mg/m²) and cisplatin (75 mg/m²) or carboplatin (AUC = 5) every 3 weeks. Patients with hypersensitivity to solvent-based paclitaxel may receive albumin-bound paclitaxel. Chemotherapy agent selection (cisplatin vs. carboplatin) is at the discretion of the investigator based on patient clinical status and organ function.

Following neoadjuvant treatment, patients will undergo concurrent chemoradiotherapy, including weekly cisplatin (40 mg/m² for 5 weeks) or carboplatin (AUC = 2), along with pelvic external beam radiation therapy (EBRT) and brachytherapy according to institutional standards.

The primary endpoints of the study are progression-free survival (PFS) as assessed by investigators per RECIST v1.1 and objective response rate (ORR) following neoadjuvant therapy. Secondary endpoints include overall survival (OS), disease control rate (DCR), duration of response (DoR), time to response (TTR), 1-year and 3-year PFS rates, 3-year and 5-year OS rates, safety (incidence and severity of adverse events), and health-related quality of life (HRQoL) as assessed by EORTC QLQ-C30.

Exploratory objectives include the identification of predictive biomarkers that may guide the clinical use of Ivonescimab in locally advanced cervical cancer.

Patients will be followed for at least 30 days for adverse events and 90 days for serious adverse events following completion of study treatment or until the start of new anticancer therapy, whichever comes first. Immune-related adverse events will be monitored for at least 90 days regardless of subsequent treatments. Survival follow-up will occur every 3 months until study completion.

This study aims to provide evidence for a potential new sequential therapeutic strategy integrating immune checkpoint blockade into the standard management of high-risk locally advanced cervical cancer

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign the written informed consent form before any study-specific procedures.
* Female participants aged ≥18 years on the day of signing informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected survival time ≥3 months.
* Histologically confirmed diagnosis of cervical cancer.
* Histological types limited to squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma.
* No prior anti-tumor treatments (including but not limited to radiotherapy, chemotherapy, surgery, targeted therapy, and immunotherapy). Note: Lymph node dissection or biopsy for clinical staging is allowed.
* FIGO 2018 stage III-IVA cervical cancer unsuitable for curative surgery. Lymph node metastasis may be confirmed by biopsy or imaging. Imaging-based lymph node metastasis must meet: MRI/CT showing positive lymph node with short-axis diameter ≥10 mm, and ≥15 mm to be used as target lesion.
* At least one measurable lesion per RECIST v1.1 criteria.
* PD-L1 CPS score ≥1 in tumor tissue.
* Must provide tumor tissue sample before treatment (FFPE blocks or ≥5 unstained slides, preferably freshly obtained).
* Adequate organ function as per screening labs:
* Hematological (without transfusion or growth factors within 2 weeks):
* ANC ≥1.5×10⁹/L
* Platelets ≥90×10⁹/L
* Hemoglobin ≥9.0 g/dL
* Renal:
* Creatinine ≤1.5×ULN or CrCl ≥50 mL/min (≥60 mL/min if cisplatin is planned), calculated by Cockcroft-Gault:

CrCl (mL/min) = [(140 - age) × weight (kg) × 0.85] / [serum creatinine (mg/dL) × 72]

* Hepatic:
* Total bilirubin ≤1.5×ULN (≤3×ULN if Gilbert's syndrome suspected)
* AST and ALT ≤2.5×ULN
* Coagulation:
* INR ≤1.5×ULN and APTT ≤1.5×ULN (unless on anticoagulants with stable dosing)
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to first dose, and agree to use effective contraception during treatment and for at least 120 days after last dose of study drug and 180 days after chemoradiotherapy.
* Effective contraception includes hormonal contraception, IUDs, or double barrier methods. Periodic abstinence and rhythm methods are not acceptable.

Exclusion Criteria:

* Cervical cancer of non-eligible histology (e.g., neuroendocrine carcinoma, sarcoma).
* Evidence of distant metastasis, including inguinal lymph node metastasis or lymph node involvement above L1 vertebral level.
* History of total hysterectomy (removal of uterus and cervix). Subtotal hysterectomy or cornuostomy preserving the cervix is acceptable.
* Anatomical or geometric contraindications to brachytherapy.
* Active malignancies within 2 years, except for treated non-melanoma skin cancer, superficial bladder cancer, in-situ breast cancer (note: cervical carcinoma in situ history is exclusionary).
* Bilateral hydronephrosis deemed non-relievable by nephrostomy or ureteral stenting.
* Anti-tumor therapy within 2 weeks before treatment initiation (including but not limited to radiotherapy, chemotherapy, surgery, targeted therapy, immunotherapy, or immuno-co-stimulatory agents like ICOS, CD40, CD137, GITR, OX40 antibodies).
* Immunomodulatory drugs (e.g., thymosin, interferon, IL-2) within 2 weeks before treatment.
* Systemic corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressants within 2 weeks, except:
* Inhaled, ophthalmic, or topical steroids ≤10 mg/day prednisone or equivalent
* Physiologic hormone replacement ≤10 mg/day prednisone or equivalent
* Prophylactic corticosteroids for hypersensitivity (e.g., CT contrast)
* Active infections requiring systemic treatment (e.g., active TB, syphilis, systemic fungal infections), except HBV antiviral therapy.
* Severe infection within 4 weeks prior to treatment (e.g., hospitalization, sepsis, severe pneumonia).
* Major surgery or significant trauma (e.g., fractures) within 4 weeks, or planned elective major surgery. Pelvic/para-aortic lymph node dissection not exclusionary.
* Live vaccines within 4 weeks.
* Active or history of autoimmune diseases except for:
* Vitiligo, alopecia, psoriasis, or eczema not requiring systemic therapy
* Autoimmune thyroiditis requiring only stable hormone therapy
* Type I diabetes requiring only stable insulin replacement
* Any of the following cardiovascular/cerebrovascular diseases:
* MI, unstable angina, PE, aortic dissection, DVT, or arterial embolism within 6 months
* NYHA Class II or greater heart failure
* Significant arrhythmias needing long-term treatment (stable asymptomatic Afib allowed)
* Stroke (CVA) within 6 months
* LVEF <50%
* History of myocarditis or cardiomyopathy
* Known primary or secondary immunodeficiency, including HIV antibody positivity.
* Active HBV infection: HBsAg positive with HBV DNA >1000 IU/mL or >5000 copies/mL; active HCV infection.
* Exception: treated and stable HBV patients with HBV DNA ≤500 IU/mL (or ≤2500 copies/mL); cured HCV patients (HCVAb+ but HCV RNA-) allowed.
* History of or active inflammatory bowel disease (Crohn's, ulcerative colitis), diverticulitis.
* Known history of allogeneic organ or stem cell transplantation.
* Interstitial lung disease or history of non-infectious pneumonitis.
* History of severe hypersensitivity to monoclonal antibodies.
* Known contraindications to cisplatin/carboplatin or paclitaxel.
* Pregnant or breastfeeding women.
* Any condition that may interfere with the study drug's safety or efficacy evaluation as judged by the investigator (e.g., other serious illness, psychiatric disorders).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is limited to biologically female participants due to the nature of cervical cancer, which affects individuals with a cervix.
Enrollment: 42 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Assessed by RECIST v1.1 | Up to 36 months
  Progression-Free Survival is defined as the time from the start of treatment until the first documented disease progression (based on RECIST v1.1 criteria, as assessed by the investigator) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
1-Year and 3-Year Progression-Free Survival (PFS) Rate | 12 months and 36 months
  The proportion of participants who remain progression-free at 1 year and 3 years from the start of treatment, assessed by RECIST v1.1 criteria
Objective Response Rate (ORR) After Concurrent Chemoradiotherapy | Within 1 month after completion of chemoradiotherapy
  The proportion of participants achieving a complete response (CR) or partial response (PR) after completing chemoradiotherapy, assessed by RECIST v1.1.
Disease Control Rate (DCR) | Up to 3 months post-treatment
  The proportion of participants achieving CR, PR, or stable disease (SD) after completion of all protocol-defined treatment, based on RECIST v1.1.
Duration of Response (DoR) | Up to 36 months
  Time from the first documented response (CR or PR) to the time of disease progression or death.
Overall Survival (OS) | Up to 60 months
  Time from treatment initiation to death from any cause.
Safety - Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From treatment initiation through 90 days post-treatment
  Incidence, severity, and type of treatment-related adverse events and serious adverse events, graded according to CTCAE v5.0.
Health-Related Quality of Life (HRQoL) | From baseline to 6 months post-treatment
  Change from baseline in patient-reported quality of life using the EORTC QLQ-C30 instrument.

OTHER OUTCOMES:
Identification of Predictive Biomarkers for Ivonescimab Efficacy | From date of randomization to 1 month after completion of chemoradiotherapy (up to approximately 4 months total)
  To explore tumor tissue and/or blood-based biomarkers that may predict response or resistance to Ivonescimab, including but not limited to PD-L1 expression, tumor-infiltrating lymphocytes (TILs), and gene expression profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Tang, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China